CLINICAL TRIAL: NCT02897349
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Parallel Group, Efficacy and Safety Study of Linagliptin, Administered Orally Once Daily, in Combination With Insulin Therapy for 24 Weeks in Chinese Type 2 Diabetes Mellitus Patients With Insufficient Glycaemic Control
Brief Title: Linagliptin Add-on to Insulin Background Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.102
Record Dates: First submitted 2016-08-30; First posted 2016-09-13 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- linagliptin (Experimental)
  Interventions: Drug: linagliptin; Drug: background therapy
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo; Drug: background therapy

INTERVENTIONS:
Drug: placebo
  Arms: Placebo
Drug: linagliptin
  Arms: linagliptin
Drug: background therapy — insulin with or without metformin

SUMMARY:
To evaluate the efficacy and safety of linagliptin compared to placebo when added on to insulin therapy alone or in combination with metformin in Chinese patients with type 2 diabetes mellitus with insufficient glycaemic control

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of type 2 diabetes mellitus prior to informed consent.
* Chinese male or female patients who are pre-treated with insulin alone or in combination with metformin:

  * With maximum insulin dose of <= 1 unit/kg/day. Acceptable basal insulins could be insulin glargin, insulin detemir or NPH (neutral protamin hagedorn) insulin with duration of action up to 24 h; acceptable pre-mixed insulins could be preparations with 25/75 or 30/70 ratio, with once or twice daily posology only. The total insulin dose should not be changed by more than 10% of the baseline value within the 12 weeks prior to randomisation (Visit 3). Both human insulin & insulin analogue are accepted.
  * If the patient is taking metformin, stable dose (at least 1500 mg daily) must be maintained for at least 12 weeks without dose adjustments prior to randomisation (Visit 3).
* HbA1c fulfills the following criteria: >= 7.5 % to <= 10.0 % at Visit 1.
* Age >= 18 years at Visit 1.
* BMI <= 45 kg/m2 (Body Mass Index) at Visit 1.
* Women of childbearing potential must be ready and able to use highly effective methods of birth control per ICH (International Conference on Harmonisation) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

  * A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile.
  * Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
* Signed and dated written informed consent by date of Visit 1 in accordance with ICH-GCP (Good Clinical Practice) and local legislation

Exclusion criteria:

* Uncontrolled hyperglycaemic with a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast during placebo run-in and confirmed by a second measurement (not on the same day).
* Any other antidiabetic drug within 3 months prior to informed consent except those defined as background treatment via inclusion criterion 2.
* Acute coronary syndrome (non-STEMI (ST Segment Elevation Myocardial Infarction), STEMI and unstable angina pectoris), stroke or TIA (Transient ischemic attack) within 3 months prior to informed consent.
* Indication of liver disease, defined by serum levels of either ALT (Alanine aminotransferase) (SGPT (serum glutamic pyruvate transaminase )), AST (Aspartate aminotransferase) (SGOT (serum glutamic-oxaloacetic transaminase)), or alkaline phosphatase above 3 × upper limit of normal (ULN (upper limit of normal)) as determined during screening and/or run-in phase.
* Any contraindications to metformin according to the local label for those patients that enter the study with metformin therapy as provided in ISF (Investigator Site File).
* Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption.
* Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years.
* Blood dyscrasias or any disorders causing hemolysis or unstable Red Blood Cell (e.g. malaria, babesiosis, haemolytic anemia).
* Known hypersensitivity or allergy to the investigational product or its recipients.
* Treatment with anti-obesity drugs 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight.
* Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except T2DM (Type 2 diabetes mellitus).
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake in the opinion of the investigator.
* Participation in another trial with an investigational drug within 2 months prior to informed consent or previous enrolment in this trial.
* Any other clinical condition that would jeopardize patient's safety while participating in this clinical trial in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (25):
- China (25):
  - China-Japan Friendship Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - The General Hospital of Chinese People's Armed Police Forces, Beijing
  - First Hospital of Jilin University, Changchun
  - No.900 Hospital of PLA Joint Logistics Support Force, Fuzhou
  - Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - General Hospital of Jinan Military Area, Jinan
  - Nanjing First Hospital, Nanjing
  - The affiliated hospital of medicalcollege qingdao university, Qingdao
  - Centre Hospital of Putuo District, Shanghai, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Yangpu Hospital, Tongji University, Shanghai
  - Second Hospital Affiliated to Shantou Medical University, Shantou
  - Shengjing Hospital of China Medical University, Shengyang
  - Siping Central People's Hospital, Siping
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Nankai University Affiliated Hospital, Tianjin
  - The 2nd Hospital of Tianjin Medical University, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Renmin Hospital of Wuhan University, Wuhan
  - First Affiliated Hospital of Xiamen University, Xiamen
  - the first people hospital of Yue Yang, Yueyang
  - Affiliated Hospital of Jiangsu University, Zhenjiang

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double-blind, multi-centre, and placebo-controlled, parallel group study to compare linagliptin with placebo as add-on therapy to stable insulin alone (basal insulin, premixed insulin) or in combination with metformin in Chinese type 2 diabetes mellitus (T2DM) participants with insufficient glycaemic control.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be randomized to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Placebo Matching Linagliptin: Participants were administered placebo matching 5 milligram (mg) linagliptin tablet once daily per os (p.o.) for 24 weeks.
- Linagliptin: Participants were administered 5 milligram (mg) linagliptin tablet once daily per os (p.o.) for 24 weeks.
Period: Overall Study
Arm/Group | Placebo Matching Linagliptin | Linagliptin
Started (Started are randomized/ treated) | 102 | 104
Completed | 97 | 98
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 3 | 3
Not completed — Other than listed above | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS) : The TS consisted of all patients treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching Linagliptin | Linagliptin | Total
Number analyzed (Participants) | 102 | 104 | 206
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (10.6) | 60.1 (9.5) | 58.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 54 | 52 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 102 | 104 | 206
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 102 | 104 | 206
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c) After 24 Weeks of Treatment
Description: Percentage change from baseline, that is, [[(HbA1c after 24 weeks of treatment) - (HbA1c at baseline)] / (HbA1c at baseline)] *100%, where baseline refers to the last observation prior to the start of randomised study drug, including the observation prior to the placebo run-in.
Time Frame: Baseline and week 24
Population: Full analysis set (FAS) observed cases (OC): The FAS consisted of all patients randomised in the TS who had a baseline HbA1c value and at least one on-treatment HbA1c value. The FAS was the basis for the intention-to-treat (ITT) analysis.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo Matching Linagliptin | Linagliptin
Number analyzed (Participants) | 99 | 100
Percentage change | -0.20 (0.09) | -0.61 (0.09)
Statistical Analysis 1: Comparison: Placebo Matching Linagliptin vs Linagliptin; Based on Mixed-effect Model Repeated Measures (MMRM) including fixed effects treatment, week, type of insulin, and treatment by week interaction, linear covariates baseline HbA1c, baseline HbA1c by week interaction and random effect for patient. Within-patient errors are modelled by unstructured covariance matrix. Adjusted mean is based on all patients in the model (not only patients with a baseline and week 24 measurement); Test type: Superiority; p = 0.0016, Mixed model repeated measures; Adjusted Mean Difference (%) = -0.40, 95% CI 2-sided [-0.65 to -0.16], Standard Error of Mean 0.13

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 24 Weeks of Treatment
Description: Change from baseline in Fasting plasma glucose (FPG) after 24 weeks of treatment.
Time Frame: Baseline and week 24
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: Milligram/Decilitre (mg/dL)
Arm/Group | Placebo Matching Linagliptin | Linagliptin
Number analyzed (Participants) | 99 | 99
Milligram/Decilitre (mg/dL) | 0.7 (3.6) | -5.5 (3.6)
Statistical Analysis 1: Comparison: Placebo Matching Linagliptin vs Linagliptin; Based on MMRM including fixed effects treatment, week, type of insulin, and treatment by week interaction, linear covariates baseline HbA1c, baseline FPG baseline FPG by week interaction and random effect for patient. Within-patient errors are modelled by unstructured covariance matrix. Adjusted mean is based on all patients in the model (not only patients with a baseline and week 24 measurement); Test type: Superiority; p = 0.2241, Mixed model repeated measures; Adjusted Mean Difference (mg/dL) = -6.2, 95% CI 2-sided [-16.2 to 3.8], Standard Error of Mean 5.1

3. Secondary Outcome: Change From Baseline in 2-hour (2-h) Postprandial Plasma Glucose (PPG) After 24 Weeks of Treatment
Description: Change from baseline in 2-hour (2-h) postprandial plasma glucose (PPG) after 24 weeks of treatment.
Time Frame: Baseline and week 24
Population: Meal tolerance test (MTT) (OC) set: MTT-set consisted all patients of the FAS with a valid MTT at baseline and at the end of the study. An MTT was considered valid if it had a valid FPG and a valid 2-h PPG value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Matching Linagliptin | Linagliptin
Number analyzed (Participants) | 78 | 88
mg/dL | -0.06 (5.98) | -32.01 (5.66)
Statistical Analysis 1: Comparison: Placebo Matching Linagliptin vs Linagliptin; Based on analysis of covariance (ANCOVA) model including fixed effect treatment and type of insulin, and linear covariates baseline HbA1c and baseline 2-h PPG; Test type: Superiority; p = 0.0001, ANCOVA; Adjusted Mean Difference (mg/dL) = -31.95, 95% CI 2-sided [-48.15 to -15.75], Standard Error of Mean 8.20

4. Secondary Outcome: Percentage of Participants With HbA1c on Treatment <7.0 Percentage (%) After 24 Weeks of Treatment
Description: Percentage of participants with HbA1c on treatment <7.0 percentage (%) after 24 weeks of treatment. Participants with baseline HbA1c <7.0% were excluded from the analysis.
Time Frame: 24 weeks
Population: Full analysis set (FAS) Non-completers considered as failure (NCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Matching Linagliptin | Linagliptin
Number analyzed (Participants) | 97 | 101
Percentage of participants | 8.2 | 13.9
Statistical Analysis 1: Comparison: Placebo Matching Linagliptin vs Linagliptin; Logistic regression model with terms for treatment and type of insulin as fixed effect and continuous linear covariates baseline HbA1c; Test type: Superiority; p = 0.2431, Regression, Logistic; Odds Ratio (OR) = 1.793, 95% CI 2-sided [0.673 to 4.780]

5. Secondary Outcome: Percentage of Participants With HbA1c on Treatment < 6.5% After 24 Weeks of Treatment
Description: Percentage of participants with HbA1c on treatment < 6.5% after 24 weeks of treatment. Participants with baseline HbA1c <6.5% were excluded from the analysis.
Time Frame: 24 weeks
Population: FAS (NCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Matching Linagliptin | Linagliptin
Number analyzed (Participants) | 100 | 101
Percentage of participants | 3.0 | 4.0
Statistical Analysis 1: Comparison: Placebo Matching Linagliptin vs Linagliptin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.6235, Regression, Logistic; Odds Ratio (OR) = 1.481, 95% CI 2-sided [0.309 to 7.105]

6. Secondary Outcome: Percentage of Participants With HbA1c Lowering by at Least 0.5% After 24 Weeks of Treatment
Description: Percentage of participants with HbA1c lowering by at least 0.5% after 24 weeks of treatment.
Time Frame: 24 weeks
Population: FAS (NCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Matching Linagliptin | Linagliptin
Number analyzed (Participants) | 100 | 101
Percentage of participants | 36.0 | 55.4
Statistical Analysis 1: Comparison: Placebo Matching Linagliptin vs Linagliptin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0049, Regression, Logistic; Odds Ratio (OR) = 2.293, 95% CI 2-sided [1.286 to 4.091]

7. Secondary Outcome: Percentage of Participants With Any Investigator-defined Hypoglycaemic Adverse Event (AE) With Plasma Glucose (PG) ≤70 mg/dL
Description: Incidence of investigator-reported hypoglycaemic events confirmed by a measured blood glucose ≤70 mg/dL (≤3.9 Millimoles Per Litre (mmol/L)). Severe hypoglycaemic AE = hypoglycaemic event requiring the assistance of another person to actively administer carbohydrate, glucagon or other resuscitative actions.
Time Frame: 24 weeks
Population: Treated set (TS) : The TS consisted of all patients treated with at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Matching Linagliptin | Linagliptin
Number analyzed (Participants) | 102 | 104
Percentage of Participants | 7.8 | 10.6

8. Secondary Outcome: Percentage of Participants With Any Severe Hypoglycaemic AE
Description: Incidence of severe hypoglycaemic events (requiring active assistance by another person, or fatal). Severe hypoglycaemic AE = hypoglycaemic event requiring the assistance of another person to actively administer carbohydrate, glucagon or other resuscitative actions.
Time Frame: 24 weeks
Population: TS
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Matching Linagliptin | Linagliptin
Number analyzed (Participants) | 102 | 104
Percentage of Participants | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after the last drug administration, up to 176 days.
Arm/Group | Placebo Matching Linagliptin | Linagliptin
All-Cause Mortality (participants affected / at risk) | 1/102 | 0/104
Serious Adverse Events (participants affected / at risk) | 17/102 | 10/104
Other Adverse Events (participants affected / at risk) | 26/102 | 33/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching Linagliptin (N=102) | Linagliptin (N=104)
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Conductive deafness (Ear and labyrinth disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 1
Ophthalmoplegia (Eye disorders) | 1 | 0
Pterygium (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 2
Facial paralysis (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching Linagliptin (N=102) | Linagliptin (N=104)
Upper respiratory tract infection (Infections and infestations) | 13 | 14
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 13 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT02897349/SAP_001.pdf
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT02897349/Prot_002.pdf